CLINICAL TRIAL: NCT00522249
Title: A Study of Pegylated Alfa Interferon, Sunitinib and Tarceva in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Study of Pegylated Alfa Interferon, Sunitinib and Tarceva in Patients With Metastatic RCC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI decision
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAC IRB#0806-0132; RCC-06-101 (Other: Principal Investigator)
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: Metastatic Renal Cell Carcinoma; RCC; M3thodist; Pegylated Alfa Interferon; Sunitinib; Tarceva; Peg IFN
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Introns; peginterferon alfa-2b; Sunitinib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): One cycle of the combination therapy will be 42 days (6 weeks). All patients will receive PEG-Intron given subcutaneously on Day 1 each week. Patients will receive Sunitinib orally on Days 1-28 of each cycle. Patients will receive Tarceva orally on Days 1-42.
  Interventions: Drug: Pegylated Alfa Interferon; Drug: sunitinib; Drug: erlotinib

INTERVENTIONS:
Drug: Pegylated Alfa Interferon — Each patient will receive PEG-Intron administered subcutaneously one day per week of each 6 week cycle. The dose of PEG-Intron is determined based on the patient's weight and the dose level.
  Other Names: Intron A; PEG Intron®; PEG-Intron Redipen®
Drug: sunitinib — Patients will receive sunitinib orally as a single daily dose on Days 1-28 of each 42-day cycle. The dose will depend on the dose level.
  Other Names: Sutent®
Drug: erlotinib — Tarceva will be administered orally, 1-42 of each 42 day cycle. Dose will depend on dose level. Supplied as 150-mg, 100-mg and 25-mg strengths, white film-coated tablets for administration.
  Other Names: Tarceva®

SUMMARY:
The purpose of this study is to evaluate the combination of Pegylated Alfa Interferon (PEG-Intron), Sunitinib and Tarceva to see if this drug combination delays the disease progression of patients with metastatic Renal Cell Carcinoma. The first phase of this study will determine the best dose of Peg-Intron, Sunitinib and Tarceva when given in combination. The safety of giving these drugs in combination and response to treatment will also be examined.

DETAILED DESCRIPTION:
Over 75% of RCCs are highly vascularized tumors that overexpress a number of growth factors, including VEGF, PDGF, and bFGF. In addition, RCC tumors overexpress the receptors for these peptides. These ligands and receptors may be involved in the autocrine stimulation of tumor cell growth, or in the paracrine stimulation of neovascular or stromal fibroblast growth that supports tumor expansion. Novel treatment that specifically interrupts these signaling pathways may have significant anti-tumor activity. When taken together, these data provide a rationale for investigation of a combination therapy with PEG-Intron, Sunitinib and Tarceva for clear cell and papillary RCC patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic or unresectable RCC. Patients must have a component of conventional clear cell renal carcinoma or papillary renal carcinoma.
* No more than three prior systemic therapies of any kind for RCC including: 1) Immunotherapy (Adjuvant vaccines, Interleukin-2, Interferon-α) 2) Chemotherapy 3) Molecular targeted agents (Nexavar [Sorafenib], Bevacizumab [Avastin]) 4) Investigational therapy
* Patients with their primary tumor in place who are appropriate surgical candidates should be strongly encouraged (but not required) to undergo nephrectomy.
* Prior palliative radiotherapy in metastatic lesion(s) is permitted, provided there is at least one measurable and/or evaluable lesion(s) that has not been irradiated.
* All major surgery of any type and/or radiotherapy must be completed at least 4 weeks prior to registration. Patients must have recovered from surgery and/or radiotherapy toxicity prior to registration.
* At the time of enrollment, patients must have evidence of metastatic or unresectable disease.
* Paraffin RCC tissue blocks or unstained slides must be obtained for future chemistry staining or every effort made to obtain samples.
* Karnofsky performance status > 70%.
* Echocardiogram ejection fraction of ≥ 45%
* Age >18.
* Must meet required initial laboratory values

Exclusion Criteria:

* Patients with true chromophobe, oncocytoma, collecting duct tumor and transitional cell carcinoma are NOT eligible.
* Patients who have received small molecule epithelial growth factor inhibitors (such as Irresa, Tarceva) are excluded.
* Patients who have had prior exposure to sunitinib are excluded.
* No ongoing hemoptysis, or cerebrovascular accident within 12 months, or peripheral vascular disease with claudication on less than 1 block, or history of clinically significant bleeding, because of the potential bleeding and/or clotting risk with this combination therapy.
* No deep venous thrombosis or pulmonary embolus within 12 months of randomization and no ongoing need for full-dose oral or parenteral anticoagulation. Low dose coumadin (1 mg) for maintenance of catheter patency or daily prophylactic aspirin is allowed.
* No evidence of current central nervous system (CNS) metastases. Any imaging abnormality indicative of CNS metastases will exclude the patient from the study.
* No significant cardiovascular disease defined as congestive heart failure (New York Heart Association Class II, II or IV) angina pectoris requiring nitrate therapy, or recent myocardial infarction (within the last 6 months).
* No active ischemia on electrocardiogram.
* No patients with uncontrolled hypertension (defined as blood pressure of > 160 mmHg systolic and/or > 90 mmHg diastolic on medication).
* - Any ongoing requirement for systemic corticosteroid therapy (except replacement therapy for adrenal insufficiency) is not permitted. Topical and/or inhaled steroids are allowed.
* Patients with a pre-existing thyroid abnormality whose thyroid function cannot be maintained in the normal range by medication are ineligible.
* No uncontrolled psychiatric disorder.
* Patients with delayed healing of wounds, ulcers, and/or bone fractures are not eligible.
* Patients with a 'currently active' second malignancy other than non-melanoma skin cancers are not eligible.
* Pregnant women are excluded (negative urine or serum pregnancy test required) because of the potential for teratogenic or abortifacient effects of therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-05; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Time to progression Objective response rate | every 6 wks

SECONDARY OUTCOMES:
Overall survival | every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, DO, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Baylor College of Medicine - Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No